CLINICAL TRIAL: NCT06007924
Title: Phase II of Avutometinib (VS-6766) and Defactinib In RAF Dimer-Driven RAI-Refractory Differentiated and Anaplastic Thyroid Cancer Patients
Brief Title: A Study of Avutometinib and Defactinib in People With Thyroid Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-007; 1R01FD008181-01 (FDA)
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Cancer
Keywords: Avutometinib; Defactinib; 23-007
MeSH Terms: conditions — Thyroid Neoplasms | interventions — defactinib

STUDY DESIGN:
Intervention Model Description: This is a phase II clinical trial evaluating avutometinib in combination with defactinib in radioiodine-refractory (RAIR), recurrent and/or metastatic differentiated thyroid cancer (DTC) (Cohort A) and anaplastic thyroid cancer (ATC) (Cohort B) patients.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Radioiodine-refractory (RAIR), recurrent and/or metastatic differentiated thyroid cancer (DTC) (Experimental): Patients will be treated with avutometinib 3.2 mg twice weekly and defactinib 200 mg twice daily, both 3 weeks on/1 week off.
  Interventions: Drug: Avutometinib; Drug: Defactinib
- Anaplastic thyroid cancer (ATC) (Experimental): Patients will be treated with avutometinib 3.2 mg twice weekly and defactinib 200 mg twice daily, both 3 weeks on/1 week off.
  Interventions: Drug: Avutometinib; Drug: Defactinib

INTERVENTIONS:
Drug: Avutometinib — Avutometinib 3.2 mg twice weekly 3 weeks on/1 week off
Drug: Defactinib — Defactinib 200 mg twice daily 3 weeks on/1 week off

SUMMARY:
The researchers are doing this study to find out if the combination of avutometinib and defactinib is an effective treatment for RAF dimer-driven radioiodine-refractory differentiated thyroid cancer or anaplastic thyroid cancer. The researchers will also test whether avutometinib and defactinib is a safe treatment that causes few or mild side effects.

ELIGIBILITY:
Inclusion Criteria:

Cohort A will enroll RAIR, R/M DTC patients with RAF dimer-driven disease.

Cohort B will enroll ATC patients with RAF dimer-driven disease.

* Cohort A only: Patients must have pathologically or cytologically confirmed differentiated thyroid cancer of follicular origin (including papillary thyroid carcinoma, follicular thyroid carcinoma, hurthle cell carcinomas, poorly differentiated thyroid carcinoma and their respective variants).
* Cohort B only: Patients must have anaplastic thyroid carcinoma.
* Confirmation in a CLIA certified laboratory that one of the patient's thyroid tumors (primary tumor, recurrent tumor, or metastases) possess at least one of the following genetic alterations: RAS mutation, NF1 mutation, RET rearrangement, NTRK rearrangement, ALK rearrangement, Class 2 or 3 BRAF alterations (non-V600E/K mutations or rearrangements).
* Cohort A only: Evidence of progressive disease (e.g. presence of new or growing lesion(s) on radiologic imaging and/or new or worsening tumor-related symptoms) within 14 months of study enrollment.
* Cohort A only: Patients must have recurrent or metastatic disease not amenable to curative surgery or radiation.
* Patients with any number of prior therapies will be eligible.
* Patients must have RECIST v1.1 measurable disease.
* Age ≥ 18 years.
* ECOG performance status of 0 or 1.
* For Cohort A only: Patients must have not had recent treatment for thyroid cancer as defined as:

  * No prior RAI therapy is allowed <6 months prior to initiation of therapy on this protocol. A diagnostic study using <10 mCi of RAI is not considered RAI therapy
  * No external beam radiation therapy <1 weeks prior to initiation of therapy on this protocol.
  * No chemotherapy or targeted therapy (e.g., tyrosine kinase inhibitor) is allowed <4 weeks prior to the initiation of therapy on this protocol
* For Cohort A only: Patients must have RAI-refractory disease, defined as one of the following:

  * Total lifetime dose of radioiodine > 600 mCi
  * A tumor that is not radioiodine-avid on a diagnostic radioiodine scan performed
  * A radioiodine-avid metastatic lesion which progressed despite radioiodine treatment given 6 months or more prior to study entry in the study. There are no size limitations for the index lesions used to satisfy this entry criterion
  * The presence of at least one fluorodeoxyglucose (FDG) avid lesion.
* Patients must be able to swallow and retain orally-administered pills without any clinically significant gastrointestinal abnormalities that may alter absorption, such as malabsorption syndrome or major resection of the stomach or bowels.
* Adequate recovery from toxicities related to prior treatments to at least Grade 1 by CTCAE v 5.0. Exceptions include alopecia and peripheral neuropathy grade ≤ 2.
* Patients must have tissue from the primary tumor or metastases available for correlative studies. Either a paraffin block or at least 20 unstained slides are acceptable (30 unstained slides would be ideal). (If less than twenty unstained slides are available and a paraffin bloc is not available, the patient may be able to participate at the discretion of the investigator).
* Patients must agree to undergo two research biopsies of (a) malignant lesion(s). Tumor tissue obtained prior to study consent or treatment as part of standard of care can also be submitted in lieu of performance of the first pre-treatment biopsy if the Principal Investigator deems it to be of sufficient quantity/quality/timeliness. Patients may also be exempt from biopsy if 1) the investigator or person performing the biopsy judges that no tumor is accessible for biopsy, 2) the investigator or person performing the biopsy feels that the biopsy poses too great of a risk to the patient (including if conduct of the biopsy will result in an unacceptable delay in therapy), or 3) the patient cannot be safely removed from anti-coagulation therapy (if the anti-coagulation therapy needs to be temporarily held for the biopsy procedure). If the only tumor accessible for biopsy is also the only lesion that can be used for RECIST v1.1 response evaluation, then the patient may be exempt from biopsy. If the investigator deems a second research biopsy to be high risk after a patient has completed the first research biopsy, the patient may be exempt from the second biopsy. Biopsies of lesions that are in proximity to any vital neurovascular structures that can be considered high risk procedures will not be biopsied.
* Baseline QTc interval < 460 ms for women and ≤450 ms for men using Frederica's QT correction formula. NOTE: This criterion does not apply to patients with a right or left bundle branch block.
* Adequate cardiac function wit left ventricular ejection fraction >50% by echocardiography (ECHO) or multiple-gated acquisition (MUGA) scan.
* Screening laboratory values must meet the following criteria:

  * WBC ≥ 2000/μL
  * Neutrophils ≥ 1000/μL
  * Platelets ≥ 100 x10^3 /μL
  * Hemoglobin > 9.0 g/dL
  * AST/ALT ≤ 2.5 x ULN (of < 5x ULN in patients with liver metastases)
  * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
  * International normalized ratio (INR) < 1.5 and partial thromboplastin time (PTT) < 1.5 x ULN in the absence of anticoagulation or therapeutic levels in the presence of anticoagulation.
  * Albumin ≥ 3.0 g/dL (451 μmole/L)
  * Creatine phosphokinase (CPK) ≤ 2.5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 50 mL/min (if using the Cockcroft-Gault formula below)
  * Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL
  * Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL

Exclusion Criteria:

* Symptomatic untreated brain or leptomeningeal metastases Note: Patients with asymptomatic or treated brain or leptomeningeal metastases are allowed. Participants with symptomatic brain or leptomeningeal metastases after surgical and/org radiation therapy may be allowed with Principal Investigator approval.
* Prior therapy with a MEK 1/2 inhibitor or an inhibitor that targets Class II/Class III BRAF alterations or a FAK inhibitor (with the exception of patients who received these therapies for a defined period of time to enhance radioiodine activity).
* Patient who have had systemic investigational anti-cancer therapy within 4 weeks of the first dose of study therapy.
* Major surgery within 4 weeks (excluding placement of vascular access), minor surgery within 2 weeks, or radiotherapy within 1 week of the first dose of study drug.
* Treatment with warfarin. Patients on warfarin for deep vein thrombosis/pulmonary embolism should be converted to low-molecular-weight heparin (LMWH) or direct oral anticoagulants (DOACs).
* Concomitant use of strong inhibitors and inducers of CYP3A4 (see Appendix 1 in Section 18). Patients should refrain from consumption of grapefruit, grapefruit juice and St. John's Wort, and other medications (with or without prescriptions), supplements, herbal remedies or foods that are strong inhibitors or inducers of CYP3A4 during treatment
* Concomitant use of strong CYP2C9 inhibtors or inducers. For additional guidance see https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-druginteractions-table-substrates-inhibitors-and-inducers
* Concomitant use of strong P-glycoprotein(P-gp) inhibitors or inducers. For additional guidance see https://www.uptodate.com/contents/image/print?imageKey=EM%2F73326&topicKey=HEME%2F1370&source=outlinelink
* Patients with history of glaucoma, history of retinal vein occlusion (RVO), predisposing factors for RVO, including uncontrolled hypertension, uncontrolled diabetes.
* Patients with a history of retinal pathology or evidence of visible retinal pathology that is considered a risk factor for RVO, such as an intraocular pressure > 21 mmHg
* Treatment-refractory hypertension defined as a blood pressure of systolic >140 mmHg and/or diastolic >90 mmHg which cannot be controlled by anti-hypertensive therapy.
* Patients with active hepatitis B infection (HBV surface antigen positive).
* Subject is known to be positive for Human Immunodeficiency Virus (HIV) or active Hepatitis C Virus (HCV). Testing for HIV or Hepatitis C prior to initiation of the study drug is not required. If a patient has a known history of treated HCV, then a viral load is required to confirm clearance of infection.
* Known severe acute respiratory syndrome coronavirus 2 SARS-Cov2 infection (clinical symptoms) ≤28 days prior to first dose of study therapy.
* History of rhabdomyolysis.
* Concurrent congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA]), myocardial infarction within the last 6 months, unstable arrhythmias, unstable angina or severe obstructive pulmonary disease.
* Subjects with the inability to swallow oral medications or impaired gastrointestinal absorption due to gastrectomy or active inflammatory bowel disease
* Any other medical condition (e.g., cardiac, gastrointestinal, pulmonary, psychiatric, neurological, genetic, etc.) that in the opinion of the Investigator places the patient at unacceptably high risk for toxicity.
* Patients who are pregnant or breastfeeding.
* Patients with hypersensitivity to mannitol, magnesium stearate, HPMC (hydroxypropyl methylcellulose) shells

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2027-08-16 (Estimated); Study Completion 2027-08-16 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) cohort A | up to 2 years
  Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)
overall response rate (ORR) cohort B | up to 2 years
  Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ho, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York
  - Lehigh Valley Health Network (Data Collection Only), Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm